CLINICAL TRIAL: NCT07062783
Title: The Effect of Respiratory and Aerobic Exercises on Neuroprotective and Inflammation Biomarkers in Patients Diagnosed With Major Depression
Brief Title: Effect of Aerobic Exercise on Biomarkers in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Scientific Research Projects Coordination Unit (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAE1
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-05

CONDITIONS: Major Depression
Keywords: Depression; Aerobic exercise; Oxidative stress; Growth factors
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Breathing Exercises; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Those included in the experimental group continued diaphragmatic breathing exercises every day for three weeks and walking exercises at least three days a week.
  Interventions: Other: Breathing exercise; Other: Aerobic Exercise
- Control group (No Intervention): The control group continued their routine lives, and at the end of three weeks

INTERVENTIONS:
Other: Breathing exercise — Volunteers participating in the study who were included in the experimental group performed breathing exercises every day for three weeks. They were taught to focus their attention on the hand on their abdominal area while breathing slowly through their nose and to increase abdominal movement while reducing chest movement. They were warned that during inspiration, as air filled their lungs, the hand on their abdomen should rise upward and the hand on their chest should not move excessively. Participants continued the training until they performed the exercise correctly. The diaphragmatic breathing exercise was performed for 10 minutes in the supine position during the first week, in the semi-sitting and/or sitting position during the second week, and in the standing position during the final week.
  Arms: Exercise Group
Other: Aerobic Exercise — The ratios determined as reference values for walking training in healthy adults (reference value for women = (2.11*height) - (2.29*body weight) - (5.78*age) + 667 meters - reference value for men = (7.57*height) - (1.76*body weight) - (5.0 2*age) - 309 meters) was performed at 80% intensity for at least 30 minutes on at least 3 days a week for 3 weeks. Aerobic exercise was considered for 3 weeks to facilitate adaptation to exercise and sustainability.
  Arms: Exercise Group

SUMMARY:
This study aims to investigate changes in the levels of biomarkers (IGF-1, FGF2, and EGF) involved in neuron development in patients diagnosed with major depression through the effects of breathing exercises and aerobic exercise, as well as to examine the levels of biomarkers (TNF-α, IL-6, and IL-1) and oxidative stress (TAS, TOS, MDA, and F2-isoprostane) that are thought to play a role in the pathophysiology of depression.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who volunteer to participate in the study,
* Between the ages of 18 and 40,
* Have been diagnosed with clinical depression by a psychiatrist according to DSM-5 criteria

Exclusion Criteria:

* Individuals with chronic conditions accompanying depression,
* Those with walking difficulties
* Those with respiratory system disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress biomarkers | From enrollment to the end of treatment at 3 weeks
  It has been reported that the interaction between oxidative stress and the immune system is important, and that activated immune inflammatory pathways can trigger oxidative stress. In our study, an ELISA test will be conducted to investigate how exercise affects the levels of oxidative stress (TAS, TOS, MDA, and F2-isoprostane) biomarkers, which play a role in the pathophysiology of depression.
Proinflmatuar sytokines | From enrollment to the end of treatment at 3 weeks
  It is believed that increased production of key proinflammatory cytokines such as interleukin tumor necrosis factor-alpha (TNF-alpha), interleukin-6 (IL-6), and interleukin-1 (IL-1) and acute phase reactants plays an important role in the development of depression as a result of immune system involvement.
  In our study, an ELISA test will be conducted to investigate how exercise affects the levels of inflammation (TNF-α, IL-6, IL-1) which play a role in the pathophysiology of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No